CLINICAL TRIAL: NCT03557073
Title: The Effects of Postoperative Physician Phone Calls for Hand and Wrist Fractures: a Single-blinded, Prospective, Randomized Controlled Trial
Brief Title: The Effects of Postoperative Physician Phone Calls for Hand and Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Joshua Adkinson, Joshua Michael Adkinson, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1712309601
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Hand Injuries; Trauma; Hand Injuries and Disorders
Keywords: Hand injuries; Hand trauma; Patient reported outcomes
MeSH Terms: conditions — Hand Injuries; Wounds and Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receiving a postoperative phone call or not receiving a postoperative phone call by a physician.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Both the provider and the outcomes assessor are blinded to participant's study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Call (Experimental): Subjects in this study arm receive a post-operative phone call by a physician.
  Interventions: Behavioral: Postoperative phone call
- No Phone call (No Intervention): Subjects in this study arm do not receive an additional post-operative phone call by a physician.

INTERVENTIONS:
Behavioral: Postoperative phone call — The intervention is a phone call on the day following surgery.
  Arms: Phone Call

SUMMARY:
This study seeks to determine if postoperative phone calls by a physician affect outcomes in hand surgery.

DETAILED DESCRIPTION:
This study seeks to determine if postoperative phone calls by a physician affect outcomes in hand surgery. Patients who require operative treatment of hand and wrist fractures are randomly assigned to a group that receives a postoperative phone call or the control group that receives the standard postoperative care. Patient reported and medical outcomes are observed starting at 1 month postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated injuries of the hand who present to a specific level 1 trauma center in the Midwestern United States
* Patients who have planned surgical treatment by a pre-specified group of surgeons

Exclusion Criteria:

* Patients who have significant trauma to other organ systems proximal to the wrist
* Patients who have open ("compound") fractures (i.e., bone is exposed)
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Brief Michigan Hand Questionnaire Score Difference | 1 month postoperatively.
  A patient reported measure of hand function on a scale of 1 to 100. 100 indicates better hand function and 1 indicates worse hand function. The measure is obtained form a survey that has been published in multiple peer reviewed articles. This score can be subtracted from preoperative score to obtain a difference in score of preoperative compared to postoperative.

OTHER OUTCOMES:
Patient compliance with treatment recommendations | 1 month postoperatively
  Patient compliance with treatment as documented in their medical record. Patients are either compliant or not compliant (values can be 0 or 1), i.e., their physician states that they followed instructions or they did not.
Patient satisfaction with their overall care | 1 month postoperatively.
  Patient satisfaction with their overall care, as determined on a 5 point Likert scale. 1 is strongly satisfied whereas 5 is strongly dissatisfied.
Patient complication | 1 month postoperatively
  Patient either has a complication or does not (values can be 0 or 1), i.e., their physician states that they had a complication.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Adkinson, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided